CLINICAL TRIAL: NCT01508364
Title: NEXTAR - NEXavar® as First TARgeted Treatment for Patients With Advanced Renal Cell Carcinoma
Brief Title: Nexavar as First Targeted Therapy in Patients With Advanced Renal Cell Carcinoma
Acronym: NEXTAR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16091; NX1111 (Other: company internal)
Record Dates: First submitted 2012-01-03; First posted 2012-01-12 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal cell carcinoma, first targeted therapy, observational study
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY 43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY 43-9006) — Dosage according to label or at discretion of the attending physician

SUMMARY:
This is an observational study which will investigate the use of Nexavar as first targeted therapy in patients with advanced renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of advanced Renal cell carcinoma (RCC) for whom the decision has been taken by the investigator to prescribe Nexavar.
* Patients who failed cytokine therapy or who are not suitable for cytokines for whom Nexavar is the first targeted drug treatment.

Exclusion Criteria:

* Prior targeted therapy for RCC
* Contraindications of Nexavar described in the Summary of Product Characteristics (SPC).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with metastatic/advanced RCC (all histologies), who failed prior cytokine therapy or are not suitable for cytokine therapy and for whom Nexavar constitutes first targeted therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of Nexavar treatment | up to 3 years

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 - 1.5 years after LPLV
Health related quality of life (HRQoL) | up to 3 years
Progression-free survival (PFS) | up to 3 years
Tumor status, of patients will be evaluated according to the categories "Complete Response", "Partial Response", "Stable Disease", "Clinical Progression", "Radiological Progression". | up to 3 years
Incidence of Treatment-emergent Adverse Events (TEAE) | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany